CLINICAL TRIAL: NCT00650104
Title: 101648/196: A Long-Term, Open-Label Continuation Study of Once Daily Administration of Ropinirole CR Tablets to Patients With Parkinson's Disease Who Completed the Previous Ropinirole CR Studies 167 or 164
Brief Title: Long-term Extension Study Evaluating Extended Release Ropinirole XL (Formerly Referred to as Ropinirole CR) in Patients Who Already Completed Either Study 167 or 164
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101468/196
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Results first posted 2010-04-21 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-04

CONDITIONS: Parkinson Disease
Keywords: ropinirole IR; efficacy; safety; open-label; long term safety; REQUIP; ropinirole XL; ropinirole CR; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Active Comparator): Open label medication - Ropinirole CR
  Interventions: Drug: Ropinirole XL (formerly CR)

INTERVENTIONS:
Drug: Ropinirole XL (formerly CR) — Active Ropinirole CR tablets of 2.0mg, 4.0mg, 8.0mg where subjects can tritrate to an stable optimum dose level of either 2.0mg, 4.0mg, 6.0mg, 8.0mg, 12mg, 16mg, 20mg, or 24mg per day.

SUMMARY:
The purpose of this study is to obtain information on the long-term safety, tolerability, and therapeutic benefit of extended release ropinirole XL, and to provide a mechanism for patients who participated in either Study 167 or Study 164 to continue receiving ropinirole XL if they chose to do so.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant/non-breast feeding females
* At least 30 years of age
* Diagnosis of idiopathic Parkinson''s disease (Hoehn & Yahr criteria)
* Completed either Study 167 or Study 164

Exclusion Criteria:

* Presence of uncontrolled psychiatric, hematological, renal, hepatic,endocrinological, neurological, cardiovascular disease or active malignancy
* Dizziness or fainting due to orthostatic hypotension on standing
* Significant sleep disorder
* Drug abuse or alcoholism

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2002-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (10):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Houston, Texas

REFERENCES:
- [Background] Hauser RA, Reichmann H, Lew M, Asgharian A, Makumi C, Shulman KJ. Long-term, open-label study of once-daily ropinirole prolonged release in early Parkinson's disease. Int J Neurosci. 2011 May;121(5):246-53. doi: 10.3109/00207454.2010.546538. Epub 2011 Jan 19. PMID 21244307

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study 101468/196 (this study; NCT#00650104) was an open-label, ropinirole XL (2-24 mg/day), continuation study for participants with Parkinson's Disease who previously completed Studies 167 or 164. Treatment was originally designed to continue for 3 years, but it was extended until ropinirole XL became commercially available in each study country.
Groups:
- Ropinirole XL: Up-titration: some participants from Study 167 started at 2 milligrams (mg) ropinirole XL once daily. Then, depending on the response/tolerance of each participant, the dose was increased in 1 mg weekly increments to 4 mg, then 2 mg weekly increments up to 12 mg, and in either 2 mg or 4 mg weekly increments up to 24 mg to the clinical optimum dose. Other Study 167 participants were increased in 2 mg weekly increments up to 8 mg and then 4 mg weekly increments up to 24 mg. Study 164 particiapnts who were on an optimal dose of ropinirole XL could go straight into the long-term treatment period, and those who were receiving ropinirole IR could be switched to the corresponding XL dose. Long-term treatment: participants received study medication until market availability of ropinirole XL. After market availability, participants would undergo a 1-week down-titration period; after protocol amendment #4 approval, participants could switch directly to the market-available dose.
Period: Overall Study
Arm/Group | Ropinirole XL
Started | 83
Completed | 42
Not Completed | 41
Not completed — Adverse Event | 17
Not completed — Death | 2
Not completed — Withdrawal by Subject | 11
Not completed — Physician Decision | 7
Not completed — Lost to Follow-up | 1
Not completed — Non-compliance | 2
Not completed — Sponsor Terminated Dosing | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 83
Age Continuous [Mean (Standard Deviation); unit: years] | 65.1 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 46
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 74
  Hispanic | 6
  Black | 1
  Asian | 1
  Other | 1
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Weight was captured during collection of demography data at baseline.
  kilograms (kg) | 79.24 (16.8)

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease (PD) Rating Scale (UPDRS) Total Activities of Daily Living Scores (Intent-to-Treat Population)
Description: The UPDRS is a clinician-based scale used to assess the longitudinal course of PD. Two of the six sections were assessed (Part II, Activities of Daily Living (ADL); Part III, Motor Examination). Both consist of a number of items (ADL, 13 items; Motor Exam., 17 items), and each item has a choice of 5 responses that are numerically scored 0-4, with 0 as the least severe response and 4 as the most severe response. ADL final score is a sum of the 13 items and may have a value between 0 (no impairment of overall activities) and 52 (severe impairment of overall activities). LTT, long-term treatment.
Time Frame: Screening; Week 4; Months 3, 9, 15, 21, 27, 33, 39, 45, 51, 57, 63, 69, 75, and 78
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study medication and who had at least one treatment period evaluation for any parameter were included in the evaluation of the therapeutic benefit. Various "n" values are the result of participant attrition.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 83
points on a scale
  Screening, n=83 | 9.4 (5.14)
  Up-titration (Week 4), n=64 | 8.9 (4.60)
  LTT, Month 3, n=76 | 8.2 (5.34)
  LTT, Month 9, n=72 | 8.1 (5.03)
  LTT, Month 15, n=67 | 9.0 (5.83)
  LTT, Month 21, n=63 | 8.6 (5.01)
  LTT, Month 27, n=58 | 9.3 (5.59)
  LTT, Month 33, n=53 | 10.3 (6.14)
  LTT, Month 39, n=19 | 10.5 (6.74)
  LTT, Month 45, n=18 | 9.3 (4.47)
  LTT, Month 51, n=19 | 10.1 (6.07)
  LTT, Month 57, n=20 | 10.4 (5.80)
  LTT, Month 63, n=19 | 11.9 (7.23)
  LTT, Month 69, n=20 | 10.8 (6.70)
  LTT, Month 75, n=16 | 12.6 (6.66)
  LTT, Month 78, n=13 | 11.5 (6.64)

2. Primary Outcome: Number of Participants With the Indicated Number of Adverse Events (AEs)
Description: AEs, defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, were collected to obtain data on the safety, tolerability, and benefit of ropinirole XL. Serious Adverse Events (SAEs), defined as AEs that are either fatal, life threatening, disabling/incapacitating, resulting in hospitalization or prolongation of a hospital stay, a congenital abnormality/birth defect, or any important medical occurrence that the investigator regards as serious based on medical judgment, were also collected. st. med., study medication.
Time Frame: Every study visit from baseline to market availability (Month 78)
Population: All participants who received at least one dose of study medication. The treatment-emergent Study 196 AEs were defined as occurring during "initial titration" or "long-term treatment" or "follow up".
Measure: Number; unit: participants
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 83
participants
  Participants (Par.) with at least one event | 81
  Par. with 0 events | 2
  Par. with 1 event | 1
  Par. with 2 events | 0
  Par. with ≥3 events | 80
  Par. with mild AEs (by maximum intensity) | 3
  Par. with moderate AEs (by maximum intensity) | 38
  Par. with severe AEs (by maximum intensity) | 40
  Par. with AEs not related to st. med. | 6
  Par. with AEs not likely related to st. med. | 6
  Par. with AEs suspected to be related to st. med. | 36
  Par. with AEs probably related to st. med. | 33
  Par. who withdrew study due to AEs | 20
  Par. reporting SAEs | 35

3. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Total Activities of Daily Living Score (Responder Population)
Description: as for outcome 1
Time Frame: Screening; Months 3, 9, 15, 27, and 78
Population: Responder: a subset of the ITT Population containing those participants who had a score of 1 (very much improved) or 2 (much improved) on the clinical global impression (CGI) scale during the study. CGI-I scores (1 to 7 [very much worse]) the participant's condition relative to baseline. Various "n" values are the result of participant attrition.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 60
points on a scale
  Screening, n=60 | 9.1 (5.08)
  LTT, Month 3, n=59 | 8.0 (5.18)
  LTT, Month 9, n=58 | 7.8 (4.92)
  LTT, Month 15, n=55 | 8.7 (5.76)
  LTT, Month 27, n=47 | 8.8 (5.80)
  LTT, Month 78, n=13 | 11.5 (6.64)

4. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Total Activities of Daily Living Scores (Maintained Responder Population)
Description: as for outcome 1
Time Frame: Screening; Months 3, 9, 15, 27, and 78
Population: Maintained Responder : subset of the Responder Population, which was maintained or further decreased for a minimum of 4 weeks whilst the participant received a stable or decreasing dose of study medication. Various "n" values are the result of participant attrition.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 47
points on a scale
  Screening, n=47 | 9.0 (5.33)
  LTT, Month 3, n=46 | 7.7 (5.53)
  LTT, Month 9, n= 46 | 7.7 (5.09)
  LTT, Month 15, n=44 | 8.6 (5.97)
  LTT, Month 27, n=37 | 8.4 (5.68)
  LTT, Month 78, n=13 | 11.5 (6.64)

5. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Motor Examination Score (ITT Population)
Description: Two of the six UPDRS sections (Part II, Activities of Daily Living (ADL); Part III, Motor Examination) were assessed in this study. The Motor Exam has 17 items, some of which are assessed in both the left and right extremities. Each item has a choice of 5 responses that are numerically scored 0-4 (0 as the least severe, 4 as the most severe). The final score is a sum of the 17 items, with some sections requiring multiple grades assigned to each extremity, and has a value ranging from 0 (no motor impairment) to 108 (severe motor impairment).
Time Frame: Screening and Month 78
Population: Intent-to-Treat (ITT) Population. Various "n" values are the result of participant attrition.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 83
points on a scale
  Screening, n=83 | 22.0 (10.14)
  Month 78, n=13 | 20.7 (7.09)

6. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Motor Examination Score (Reponder Population)
Description: as for outcome 5
Time Frame: Screening and Month 78
Population: Responder Population. Various "n" values are the result of participant attrition.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 60
points on a scale
  Screening, n=60 | 21.7 (9.71)
  Month 78, n=13 | 20.7 (7.09)

7. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Motor Examination Score (Maintained Responder Population)
Description: as for outcome 5
Time Frame: Screening and Month 78
Population: Maintained Responder Population. Various "n" values are the result of participant attrition.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 47
points on a scale
  Screening, n=47 | 22.2 (10.11)
  Month 78, n=13 | 20.7 (7.09)

8. Secondary Outcome: Number of Participants With the Indicated Responses for CGI Global Impression (CGI-I) (ITT Population)
Description: The Clinical Global Impression (CGI) scale comprises the following three components (CGI-Severity, CGI-Improvement, Index); where only the CGI-S and CGI-I were assessed in this study. CGI-I is a global improvement scale that scores the clinician's view of the participant's global functioning prior to and after initiating a study medication from 1 (very much improved) to 7 (very much worse). 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse.
Time Frame: Week 2, Month 12, Month 78
Population: Intent-to-Treat (ITT) Population. Various "n" values are the result of participant attrition.
Measure: Number; unit: participants
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 70
participants
  Week 2 - Very Much Improved, n=70 | 0
  Week 2 - Much Improved, n=70 | 2
  Week 2 - Minimally Improved, n=70 | 20
  Week 2 - No Change, n=70 | 43
  Week 2 - Minimally Worse, n=70 | 4
  Week 2 - Much Worse, n=70 | 1
  Week 2 - Very Much Worse, n=70 | 0
  Month 12 - Very Much Improved, n=69 | 7
  Month 12 - Much Improved, n=69 | 25
  Month 12 - Minimally Improved, n=69 | 20
  Month 12 - No Change, n=69 | 7
  Month 12 - Minimally Worse, n=69 | 8
  Month 12 - Much Worse, n=69 | 1
  Month 12 - Very Much Worse, n=69 | 0
  Month 78 -Very Much Improved, n=13 | 1
  Month 78 - Much Improved, n=13 | 8
  Month 78 - Minimally Improved, n=13 | 1
  Month 78 - No Change, n=13 | 1
  Month 78 - Minimally Worse, n=13 | 1
  Month 78 - Much Worse, n=13 | 0
  Month 78 - Very Much Worse, n=13 | 0

9. Secondary Outcome: Number of Participants With the Indicated Responses for CGI Global Impression (CGI-I) (Responder Population)
Description: as for outcome 8
Time Frame: Week 2, Month 12, Month 78
Population: Responder Population. Various "n" values are the result of participant attrition.
Measure: Number; unit: participants
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 56
participants
  Week 2 - Very Much Improved, n=49 | 0
  Week 2 - Much Improved, n=49 | 2
  Week 2 - Minimally Improved, n=49 | 17
  Week 2 - No Change, n=49 | 27
  Week 2 - Minimally Worse, n=49 | 2
  Week 2 - Much Worse, n=49 | 1
  Week 2 - Very Much Worse, n=49 | 0
  Month 12 - Very Much Improved, n=56 | 7
  Month 12 - Much Improved, n=56 | 25
  Month 12 - Minimally Improved, n=56 | 12
  Month 12 - No Change, n=56 | 5
  Month 12 - Minimally Worse, n=56 | 5
  Month 12 - Much Worse, n=56 | 1
  Month 12 - Very Much Worse, n=56 | 0
  Month 78 - Very Much Improved, n=13 | 1
  Month 78 - Much Improved, n=13 | 8
  Month 78 - Minimally Improved, n=13 | 1
  Month 78 - No Change, n=13 | 1
  Month 78 - Minimally Worse, n=13 | 1
  Month 78 - Much Worse, n=13 | 0
  Month 78 - Very Much Worse, n=13 | 0

10. Secondary Outcome: Number of Participants With the Indicated Responses for CGI Global Impression (CGI-I) (Maintained Responder Population)
Description: as for outcome 8
Time Frame: Week 2, Month 12, Month 78
Population: Maintained Responder Population. Various "n" values are the result of participant attrition.
Measure: Number; unit: participants
Arm/Group | Ropinirole XL
Number analyzed (Participants) | 46
participants
  Week 2 - Very Much Improved, n=37 | 0
  Week 2 - Much Improved, n=37 | 2
  Week 2 - Minimally Improved, n=37 | 12
  Week 2 - No Change, n=37 | 20
  Week 2 - Minimally Worse, n=37 | 2
  Week 2 - Much Worse, n=37 | 1
  Week 2 - Very Much Worse, n=37 | 0
  Month 12 - Very Much Improved, n=46 | 6
  Month 12 - Much Improved, n=46 | 23
  Month 12 - Minimally Improved, n=46 | 7
  Month 12 - No Change, n=46 | 4
  Month 12 - Minimally Worse, n=46 | 4
  Month 12 - Much Worse, n=46 | 1
  Month 12 - Very Much Worse, n=46 | 0
  Month 78 - Very Much Improved, n=13 | 1
  Month 78 - Much Improved, n=13 | 8
  Month 78 - Minimally Improved, n=13 | 1
  Month 78 - No Change, n=13 | 1
  Month 78 - Minimally Worse, n=13 | 1
  Month 78 - Much Worse, n=13 | 0
  Month 78 - Very Much Worse, n=13 | 0

ADVERSE EVENTS:
Time Frame: On therapy adverse events (AEs) were defined as occurring after administration of the first dose of study medication and on or before the final visit. AEs were reviewed and recorded at every visit.
Arm/Group | Ropinirole XL
Serious Adverse Events (participants affected / at risk) | 34/83
Other Adverse Events (participants affected / at risk) | 83/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole XL (N=83)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Chest pain (General disorders) | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Non-cardiac chest pain (General disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Coronary heart disease (Cardiac disorders) | 2
Overdose (Injury, poisoning and procedural complications) | 2
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 2
Muscle strain (Musculoskeletal and connective tissue disorders) | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 2
Femoral neck fracture (Musculoskeletal and connective tissue disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Delirium (Psychiatric disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Appendiceal abcess (Infections and infestations) | 1
Encephalopathy (Nervous system disorders) | 1
Postoperative wound infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastritis (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Atrial flutter (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Bronchial irritiation (Respiratory, thoracic and mediastinal disorders) | 1
Tracheobronchitis (Infections and infestations) | 1
Biliary colic (Hepatobiliary disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Spondylisthesis (Musculoskeletal and connective tissue disorders) | 1
Postoerative ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Delusion (Psychiatric disorders) | 1
Paranoia (Psychiatric disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Obsessive-complusive disorder (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Oedema peripheral (General disorders) | 1
Syncope (Nervous system disorders) | 1
Urosepsis (Infections and infestations) | 1
Accident (Injury, poisoning and procedural complications) | 1
Aortic aneurysm rupture (Blood and lymphatic system disorders) | 1
Malaise (General disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole XL (N=83)
Nausea (Gastrointestinal disorders) | 35
Dizziness (Nervous system disorders) | 34
Oedema peripheral (General disorders) | 32
Back pain (Musculoskeletal and connective tissue disorders) | 28
Headache (Nervous system disorders) | 26
Nasopharyngitis (Infections and infestations) | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 23
Somnolence (Nervous system disorders) | 23
Insomnia (Psychiatric disorders) | 22
Constipation (Gastrointestinal disorders) | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Fatigue (General disorders) | 20
Diarrhoea (Gastrointestinal disorders) | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19
Depression (Psychiatric disorders) | 18
Upper respiratory tract infection (Infections and infestations) | 15
Vomiting (Gastrointestinal disorders) | 15
Hallucination (Psychiatric disorders) | 14
Fall (Injury, poisoning and procedural complications) | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Bronchitis (Infections and infestations) | 12
Hypoaesthesia (Nervous system disorders) | 12
Tremor (Nervous system disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 12
Anxiety (Psychiatric disorders) | 12
Confusional state (Psychiatric disorders) | 11
Urinary tract infection (Infections and infestations) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10
Vision blurred (Eye disorders) | 10
Gastrointestinal reflux disease (Gastrointestinal disorders) | 10
Tooth infection (Infections and infestations) | 9
Asthenia (General disorders) | 9
Hypertension (Blood and lymphatic system disorders) | 9
Balance disorder (Nervous system disorders) | 6
Cognitive disorder (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 5
Parkinson's disease (Nervous system disorders) | 5
Sinus headache (Nervous system disorders) | 5
Dry mouth (Gastrointestinal disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 5
Joint swelling (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Flatulence (Gastrointestinal disorders) | 5
Influenza (Infections and infestations) | 7
Herpes zoster (Infections and infestations) | 5
Chest pain (General disorders) | 7
Pain (General disorders) | 6
Nightmare (Psychiatric disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Muscle strain (Injury, poisoning and procedural complications) | 5
Rash (Skin and subcutaneous tissue disorders) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5
Cataract (Eye disorders) | 5
Weight decreased (Investigations) | 5
Orthostatic hypotension (Blood and lymphatic system disorders) | 7
Angina pectoris (Cardiac disorders) | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.